CLINICAL TRIAL: NCT01542853
Title: Preliminary Study. The Value of 18F-FDG PET/CT Compared to MRI in Diagnosing Residual Disease in Patients With Spondylodiscitis
Brief Title: The Value of PET/CT in Diagnosing Residual Disease in Patients With Spinal Infection
Status: Suspended | Type: Observational
Why Stopped: problems with recruitment and funding
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Michala Kehrer, MD, MD, Odense University Hospital
Other Study IDs: spondylodiscitis-pilot
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Spondylodiscitis
MeSH Terms: conditions — Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood

SUMMARY:
MRI has shoved little correlation with the clinical finding during treatment of spondylodiscitis (infection in the vertebrae and/or discs). Since PET/CT is almost as good as MRI in diagnosing spondylodiscitis the hypothesis and this study is that PET/CT is better in predicting residual disease in patients with spondylodiscitis.

Preliminary study.

DETAILED DESCRIPTION:
In the last years there has been reported increasing incidence of spondylodiscitis. The increase is mainly thought to be caused by the increasing elderly population and the increasing amount of spinal instrumentation in this population. The symptoms range from backache to severe neurological deficits. Up to 1/3 of cases are reported to be culture negative and cases can therefore be difficult to diagnose.

MRI is thought to be the main imaging technique to visualise infection. But with the increasing availability of 18-F FDG PET/CT, it is reported to be nearly as efficient to diagnose spinal infection.

During the long antibiotic treatment of spondylodiscitis, the clinicians have no real good imaging technique to predict residual disease since MRI during the remodelling fase of the spine will mimic no difference or worsening.

Since 18-F-FDG PET marks areas with a high amount of inflammatory cells it may also be faster in returning to normal images and therefore correlates better to actual status than MRI.

Some of the purposes of this study are therefore:

* To describe changes on PET/CT and MRI at index and after 4, 8 12 and 26 weeks and compare these to the clinical findings as well as inflammatory biomarkers.
* To investigate the correlation between normalisation of inflammatory biomarkers and changes on MRI and PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* first case of infectious spondylodiscitis
* MRI or 18-F-FDG PET/CT compatible with spondylodiscitis
* overall assessment compatible with spondylodiscitis

Exclusion Criteria:

* previous spinal infection (e.g. spondylodiscitis; epidural abscess)
* spinal operation in the previous 6 months
* spinal foreign body
* current malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with MRI or PET/CT findings as well as overall clinical assessment compatible with spondylodiscitis.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-03; Study Completion 2013-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Court Pedersen, MD, DMSc, Study Chair — department of infectious diseases, Odense University Hospital; michala Kehrer, MD, Principal Investigator — Department of infectious diseases, Odense University Hospital, Denmark
Locations (3):
- Denmark (3):
  - department of nuclear medicine, Odense University Hospital, Odense
  - Department of radiology, Odense University Hospital, Odense
  - Department of infectious diseases, Odense University Hospital, Odense C